CLINICAL TRIAL: NCT00841854
Title: Comparison of 7-day and 14-day Bismuth Based Quadruple Therapy for Secondary Helicobacter Pylori Eradication.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Asan Medical Center (Other)
Collaborators: Inje University (Other); Pacific Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Hwoon-Yong Jung, M.D., Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2008-0088
Record Dates: First submitted 2009-02-10; First posted 2009-02-11 (Estimated); Last update posted 2016-12-06 (Estimated); Status verified 2016-12

CONDITIONS: Helicobacter Infection
Keywords: Helicobacter pylori; Bismuth; Salvage treatment; Metronidazole
MeSH Terms: conditions — Helicobacter Infections | interventions — Pantoprazole; Bismuth; Metronidazole; Tetracycline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- PBMT7 (Active Comparator): pantoprazole 40mg bid, bismuth 300mg qid, metronidazole 500mg tid,tetracycline 500mg qid for 7 days
  Interventions: Drug: pantoprazole; Drug: bismuth; Drug: metronidazole; Drug: tetracycline
- PBMT14 (Active Comparator): pantoprazole 40mg bid, bismuth 300mg qid, metronidazole 500mg tid,tetracycline 500mg qid for 14 days
  Interventions: Drug: pantoprazole; Drug: bismuth; Drug: metronidazole; Drug: tetracycline

INTERVENTIONS:
Drug: pantoprazole — pantoprazole 40mg bid
Drug: bismuth — bismuth 300mg qid
Drug: metronidazole — metronidazole 500mg tid
Drug: tetracycline — tetracycline 500mg qid

SUMMARY:
At present, triple therapy are recommended by various guidelines for the treatment of Helicobacter pylori (H. pylori) infection. Recent studies have shown worldwide high treatment failure rates with one week first line clarithromycin based triple therapy necessitating salvage strategy to eradicate H. pylori in primary treatment failure. However, the exact duration of bismuth based second line treatment is not determined. Therefore, the investigators performed this study to evaluate the eradication rate of 1 or 2-week quadruple regimen as a second-line therapy.

ELIGIBILITY:
Inclusion Criteria:

* H. pylori infection
* Aged between 18-80 years
* Are willing to received eradication therapy for H. pylori

Exclusion Criteria:

* Children and teenagers aged less than 18 years or over 80 years
* Previous eradication therapy for H. pylori
* History of gastrectomy
* Previous allergic reaction to antibiotics
* Use of prompt pump inhibitors and antibiotics in the recent 4 weeks
* Active upper GI bleeding in the recent 1 week
* Contraindication to treatment drugs
* Pregnant or lactating women
* Severe concurrent disease or malignancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 199 (Actual)
Dates: Start 2008-06; Primary Completion 2010-05 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Whether the two week group yield a higher eradication rate comparing to the one week group. | At least four week after completion of treatment

SECONDARY OUTCOMES:
side effect | four weeks after completion of medication

CONTACTS AND LOCATIONS:
Overall Officials: Hwoon-Yong Jung, M.D, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea

REFERENCES:
- [Derived] Chung JW, Lee JH, Jung HY, Yun SC, Oh TH, Choi KD, Song HJ, Lee GH, Kim JH. Second-line Helicobacter pylori eradication: a randomized comparison of 1-week or 2-week bismuth-containing quadruple therapy. Helicobacter. 2011 Aug;16(4):289-94. doi: 10.1111/j.1523-5378.2011.00844.x. PMID 21762268